CLINICAL TRIAL: NCT04233190
Title: A Randomized, Parallel-group, Open, Two-period, Comparative Non-inferiority Study of Eurofarma's Formoterol/budesonide Vs Alenia in the Treatment of Moderate to Severe Persistent Asthma with and Without Chronic Obstructive Pulmonary COPD
Brief Title: A Multicenter, Randomized, Parallel, Two-period, Non-inferiority Study of EurofarmavsAlenia in Asthma and COPD Treatment
Acronym: ESPIRE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eurofarma Laboratorios S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EF162
Record Dates: First submitted 2020-01-15; First posted 2020-01-18 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Asthma Copd

STUDY DESIGN:
Intervention Model Description: In the first study period (Period 1), patients with moderate to severe persistent asthma according to GINA criteria, with or without COPD, will be randomized at a 1: 1 ratio to receive formoterol 12mcg / budesonide 400mcg Eurofarma or Alenia® 12mcg / 400mcg during 12 weeks Participants who maintain asthma control at the end of this treatment period (no more than one exacerbation during this period) will be included in Period 2, in which the dose of each investigational product will be reduced (step-down), and the patients will receive formoterol 6mcg / budesonide 200mcg Eurofarma or Alenia® 6mcg / 200mcg, respectively, for an additional 12 weeks. The primary non-inferiority assessment will be performed at the end of 24 weeks of treatment, with intermediate assessment at the end of week 12.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Formoterol + budesonide Eurofarma (12/400mcg e 6/200mcg) (Experimental): Formoterol 12mcg + budesonide 400mcg / Formoterol 6mcg + budesonide 200mcg
- Alenia® (12/400mcg e 6/200mcg) (Active Comparator): Alenia® 12mcg + 400mcg / Alenia® 6mcg + 200mcg
  Interventions: Drug: Alenia® 12mcg + 400mcg / Alenia® 6mcg + 200mcg

INTERVENTIONS:
Drug: Alenia® 12mcg + 400mcg / Alenia® 6mcg + 200mcg — one inhalation, twice daily
  Other Names: fumarato de formoterol di-hidratado 12mcg + budesonida 400mcg/fumarato de formoterol di-hidratado 62mcg + budesonida 200mcg
  Arms: Alenia® (12/400mcg e 6/200mcg)

SUMMARY:
A phase III study, multicenter, randomized, parallel, open, two-period, comparative non-inferiority of Eurofarma versus Alenia® in the treatment of moderate to severe persistent asthma with and without obstructive pulmonary disease (COPD).

⚠️study will only be conducted in research centers in Brazil (please do not send e-mail if your center is outside brazil).

DETAILED DESCRIPTION:
In the first study period (Period 1), patients with moderate to severe persistent asthma according to GINA criteria, with or without COPD, will be randomized at a 1: 1 ratio to receive formoterol 12mcg / budesonide 400mcg Eurofarma or Alenia® 12mcg / 400mcg during 12 weeks Participants who maintain asthma control at the end of this treatment period (no more than one exacerbation during this period) will be included in Period 2, in which the dose of each investigational product will be reduced (step-down), and the patients will receive formoterol 6mcg / budesonide 200mcg Eurofarma or Alenia® 6mcg / 200mcg, respectively, for an additional 12 weeks. The primary non-inferiority assessment will be performed at the end of 24 weeks of treatment, with intermediate assessment at the end of week 12.

The study will be conducted in an open label since the devices for inhalation of products have different aspects, making it impossible to blind the treatments of the study. The primary efficacy variable (forced expiratory volume in one second [FEV1]) minimizes the potential bias arising from the open label of the study.

⚠️study will only be conducted in research centers in Brazil (please do not send e-mail if your center is outside brazil).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 12 years
* Presence of moderate to severe persistent asthma according to Global Initiative for Asthma (GINA) 1 criteria for at least 1 year, clinically stable (controlled) for at least 30 days.

Exclusion Criteria:

* Occurrence of asthma exacerbation within 30 days prior to initiation of study treatment.
* Presence of acute or chronic symptomatic airway infection.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 472 (Actual)
Dates: Start 2023-04-19 (Actual); Primary Completion 2024-10-28 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
FEV1 | 24 weeks
  Average change from baseline in pre-dose Forced Expiratory Volume in one second

CONTACTS AND LOCATIONS:
Locations (1):
- Eurofarma Laboratorios S.A, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No